CLINICAL TRIAL: NCT05656781
Title: An Innovative Brief Intervention Contact Program to Improve Healthcare Delivery for Suicidal Behaviour
Brief Title: Brief Intervention and Contact Program Main Trial
Acronym: BIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Zainab Samaan (Zena), Principal Investigator, Associate Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14566 HAH-22-012
Record Dates: First submitted 2022-11-10; First posted 2022-12-19 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Suicidal Behavior
Keywords: suicide; thoughts; attempts; brief intervention; contact
MeSH Terms: conditions — Suicide | interventions — Crisis Intervention; imidazole mustard

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm - Brief Intervention & Contact (Experimental): Brief education about suicidal behaviour and follow up contacts for 6 months in addition to treatment as usual. follow up will occur at the following time points post discharge: weeks 1, 2, 4, 6, 8, 12, 16 and 20. this will occur in addition to treatment as usual.
  Interventions: Other: Brief Intervention and Contact (BIC) based on Word Health Organization (WHO)
- Control (No Intervention): Control will continue treatment as usual which is whatever the clinical team decides upon post discharge. Data will be collected on repeated suicidal behaviour through medical records with consent.

INTERVENTIONS:
Other: Brief Intervention and Contact (BIC) based on Word Health Organization (WHO) — Intervention based on: Clinical WHO - SUICIDE PREVENTION DOCUMENT MULTISITE INTERVENTION STUDY ON SUICIDAL BEHAVIOURS - SUPRE-MISS: PROTOCOL OF SUPRE-MISS. Brief Intervention and Contact with participants using follow up questions about mood or any suicide attempts.
  Other Names: Brief Intervention and Contact (BIC)
  Arms: Intervention Arm - Brief Intervention & Contact

SUMMARY:
Suicide is a significant public health concern and causes approximately 1.5% of all deaths in the general population in Canada. Research shows that for individuals with comorbid psychiatric illness and suicidal behaviour, the risk of further suicide attempts persists in the first two years post-discharge with the most vulnerable time being the period immediately post discharge.

Several studies have found that alongside usual treatment, follow-up with discharged patients through text messaging, phone calls and letters, contributes to a reduction in attempts and death by suicide, and instances of self-harm. In particular, brief contact interventions have shown positive impacts in reducing further completed suicide and suicidal behaviour in patients presenting to the emergency department following a suicide attempt.

The BIC model followed in this study is adapted from the WHO protocol that was utilised as part of the Multisite Intervention Study On Suicidal Behaviours (SUPRE-MISS).

DETAILED DESCRIPTION:
Rationale The time post discharge from psychiatric hospital is a vulnerable time for suicide risk especially in patients with past suicidal behaviour as they are less likely to adhere to treatment post discharge with risk of being disengaged from healthcare services. The period after discharge therefore presents as a gap in patient care that needs to be addressed. Brief contact interventions are seen as a potential solution to this gap, thus providing justification for a trial such as this one, to test the effectiveness in a Canadian population.

Significance The rate of death by suicide has been static for past 20 years however suicidal behaviour is more dynamic with variable rates seen in those identified as high risk groups including those with a history of suicidal behaviour, males, youth, and the indigenous community. As such, there is a need to identify a feasible and accessible risk reduction strategy that can mitigate suicidal behaviour and empower individuals to leverage their social support system. We have completed a feasibility and pilot RCT study of BIC in one centre including 60 participants followed up for 6 months, which demonstrates the feasibility and justification of a main trial.

Innovation This is the first RCT that aims to impact and improve healthcare service delivery for patients with suicidal behaviour by testing a pragmatic intervention that can be easily translated into regular medical practice across institutions. This RCT builds on a pilot and feasibility trial, which has allowed for quality improvements that tailor the intervention to fit seamlessly into the discharge process. Specifically,

1. A warm transfer has been incorporated into the study design to help the intervention resemble what it would look like if it were translated into regular medical practice. This warm transfer is also important as the highest loss to follow-up rates were seen in the first point of contact post-discharge. As such, a warm transfer will remind and inform the participant that they will be receiving support and contact post hospital discharge, impacting and improving healthcare service delivery.
2. The Harbinger of Hope letter drafted by a person with lived experience will be given to the participants in the intervention arm, which directly impacts and improves healthcare service delivery by considering communication and peer supports outside of the regular care team. Participants will also be notified about the BeSafe smartphone and web application to access community support services specific to their needs (i.e. peer support, housing support, crisis services etc.), further emphasizing the focus on care outside of the most resources intense healthcare team.
3. The incorporation of a unified text message and phone call system, through a major cellular service provider, combined with the mailing of resources to participants in the intervention arm, represent advanced communication and flexible contact strategies that improve patients' accessibility and delivery of healthcare. Currently using text messaging is not possible through usual hospital communications. Participants in the pilot trial identified text messages as a preferred and low-cost option for them.
4. The incorporation of a qualitative component inquiring about participants experiences with healthcare services and the intervention will encourage participants to continue to engage in the contacts that are provided to them as the open-ended questions may be cathartic and provide a space for them to express their voices. The focus on the participants' voices once again profoundly impacts and improves healthcare service delivery by providing a platform for participants to engage. This this may also reduce disengagement and "no show" rates to appointments.
5. The primary outcomes for this study include a reduction in suicidal behaviour (death by suicide, suicide attempts and thoughts) and healthcare utilization (ER visits & readmissions), and an observation of the use of crisis service calls. The occurrence of these outcomes was lower in the intervention arm compared to the control arm when assessed in the pilot and feasibility trial (figure 1.0), which provides the justification for selecting these outcomes in a larger trial. Having these synonymous, clear, and measurable outcomes for the RCT will allow for the appropriate assessment of the effectiveness of BIC and will directly inform the translation of BIC into medical practice.
6. Crisis services were alerted during two of the phone contacts in the pilot and feasibility trial due to risk of the participant engaging in a suicide attempt which was averted. This highlights the clinical significance of the pilot and feasibility trial and provides a strong basis to continue the evaluation of the BIC intervention to eventually incorporate it into regular medical practice. It also provides evidence for the improvement of healthcare delivery as these follow-ups with participants provide the opportunity for them to re-engage with mental health services when needed and provides them with more options than an emergency room visit.
7. BIC was implemented by research staff in the pilot and feasibility trial. It will continue to be performed by research assistants that have received the appropriate safety, sensitivity, and informational trainings. This provides yet another key transferable aspect of the intervention into regular medical practice as there is no requirement for the intervention to be carried out by a mental health professional and can be administered by BIC trained personnel thus reducing the demands on services and intensive training required to deliver mental health care.

OBJECTIVES

1. Our primary aims are A) to assess the effectiveness of BIC on reducing suicidal behaviour (i.e., death by suicide and suicide thoughts/ideas and attempts) and healthcare utilization (i.e., ER visits & readmissions) post hospital discharge. B) assess the effects of BIC on crisis services used post discharge
2. Our secondary aims are to use qualitative semi-structured interviews A) to understand participants' experiences with healthcare services post discharge, including descriptions of:

   1. Participants' satisfaction with healthcare services
   2. Participants' expectations of healthcare services
   3. Participants' perceived level of social connectivity and social support

B) to understand participants' experiences with the BIC intervention, including descriptions of:

1. Participants' satisfaction with the intervention
2. Participants' perspective on the effectiveness of the intervention
3. Changes participants want to make to the intervention
4. Participants' experiences with the Harbinger of Hope letter given to them during the intervention

ELIGIBILITY:
Inclusion Criteria:

* Admitted following a suicidal behaviour (suicide attempt or with suicidal ideation),
* At least 16 years of age, no restrictions on sex or gender
* Provide written, informed consent,
* Provide consent for research staff to have access to their electronic medical record (EMR),
* Provide consent for research staff to contact their primary care provider, outpatient and other healthcare providers care team, if necessary,
* Provide health card number and consent to share with Institute for Clinical Evaluative Sciences and link to Ontario health records to analyze and evaluate events such as admissions, death by suicide and usage of health care services (such as hospitalizations) in Ontario for the period covering the study time and 2 years post study completion. The 2 years post discharge will not be feasible to continue follow up for this trial and are reported to be a risk period in the literature. Therefore, we opted to leverage administrative health record data to enrich the study impact post study completion.

Exclusion criteria

- We will exclude patients who are unable to understand written and spoken English, as the research staff/clinicians delivering the intervention are limited to English-speaking populations.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Suicidal behaviour | 6 months
  Completed and attempted suicides will be measured using yes/no questions on a self-report questionnaire and will be corroborated using electronic medical record data
Healthcare service utilization | 6 months
  This outcome will be measured using a questionnaire asking if any of the following supports were contacted:
  psychiatric or general hospital, out-patient psychiatric service, policlinic service, day-care centre, community mental health care, private psychologist or psychiatrist, consultation service for alcohol and drug related problems, consultation service for relational and sexual problems, self-help group, telephone help line, relatives, friends
Crisis services | 6 months
  This outcome will be measured using electronic medical record data indicating the number of times crisis phones calls were made and the number of emergency department visits occurred.

SECONDARY OUTCOMES:
Experiences with healthcare services post discharge | 6 months
  This outcome will be assessed qualitatively by inductively drawing themes from data collected using semi-structured interviews. Interview questions will include discussions about:
  1. Participants' satisfaction with healthcare services
  2. Participants' expectations of healthcare services
  3. Participants' perceived level of social connectivity and social support
Experiences with the BIC intervention | 6 months
  Participants' satisfaction with the intervention will be assessed qualitatively by inductively drawing themes from data collected using semi-structured interviews. Interview questions will include discussions about
  * Participants' perspective on the effectiveness of the intervention
  * Changes participants want to make to the intervention
  * Participants' experiences with the Harbinger of Hope letter given to them during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Samaan, MD/PhD, Principal Investigator — McMaster Unversity
Locations (1):
- St. Joseph's Healthcare, Hamilton, Canada

IPD SHARING:
Plan to Share IPD: No